CLINICAL TRIAL: NCT00197860
Title: Vaccination With Autologous Dendritic Cells Pulsed With Tumor Antigens for Treatment of Patients With Renal Cell Carcinoma.A Phase I/II Study.
Brief Title: Dendritic Cell Based Therapy of Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UR0414
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Advanced Renal Cell Carcinoma
Keywords: dendritic cell; vaccine; renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

INTERVENTIONS:
Biological: tumor antigen loaded autologous dendritic cells — DC vaccination regime consists of primary 10 intradermal injections of 1-2 weeks interval (q1w x 4 → q2w x 6). HLA-A2 positive patients are treated with survivin and telomerase peptide-pulsed dendritic cells, and HLA-A2 negative patients are treated with allogeneic tumor lysate-pulsed dendritic cells i.d. 1,6 mg Thymosin alpha 1 (Zadaxin®, SciClone) is administered s.c. twice a week and from the 2nd vaccine, 2 MIU Interleukin-2 is administered s.c. on day 2-6.

SUMMARY:
The purpose of this study is to show if vaccination with autologous dendritic cells pulsed with peptides or tumor lysate in combination with adjuvant cytokines can induce a measurable immune response in patients with metastatic renal cell carcinoma, and to evaluate the clinical effect (objective response rate) of the vaccination regime.

DETAILED DESCRIPTION:
Eligible patients receive vaccination with tumor antigen pulsed autologous monocyte-derived mature dendritic cells with a fixed interval. The dendritic cells are generated from leukapheresis products and frozen after antigen loading.

HLA A2 positive patients are treated with PADRE and oncopeptide pulsed DC; survivin and telomerase peptides. HLA A2 negative patients are treated with KLH and tumorlysate pulsed DC; autologous or allogeneic. Each patient is given 6 immunizations with at least 5x106 peptide/lysate pulsed autologous DC. Vaccination 1-4 is given weekly and 4-6 at 2-week intervals. Those patients who exhibit stable disease, partial response or complete response after 6 injections will be given 4 more vaccinations at 2-week interval. The vaccine is applied by intradermal injection near the inguinal region. IL-2 2 MIU s.c. day 2-6 and Thymosin alpha 1 (Zadaxin®, SciClone) 1,6 mg s.c. twice a week are used for adjuvants. Scans and re-staging tests are performed at scheduled intervals throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven progressive metastatic or locally advanced renal cell carcinoma
* No standard treatment indicated
* Age: > 18
* WHO-Performance Status 0-1
* At least tone measurable tumor lesions according to the RECIST criteria.
* Life expectancy more than 3 months
* Acceptable CBC and blood chemistry results
* Written informed consent

Exclusion Criteria:

* Patients with a history of any other neoplastic disease less than 5 years ago (excepting treated carcinomas in situ of the cervix and basal/squamous cell carcinomas of the skin).
* Patients with metastatic disease in the central nervous system (CNS).
* Patients with other significant illness including severe allergy, asthma, angina pectoris or congestive heart failure.
* Patients with acute or chronic infection including HIV, hepatitis and tuberculosis.
* Patients who are pregnant.
* Patients who have received antineoplastic therapy including chemotherapy or immunotherapy less than 4 weeks before beginning the trial.
* Patients who receive corticosteroids or other immunosuppressive agents.
* Baseline serum LDH greater than 4 times the upper limit of normal.
* Patients with active autoimmune diseases such as lupus erythematosus, rheumatoid arthritis or thyroiditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-09; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Primary aim of the study is to evaluate tolerability and safety of the treatment. | weekly for the first four weeks, thereafter biweekly

SECONDARY OUTCOMES:
Secondary aims: evaluation of treatment induced immune response and clinical response. | after 8 and 16 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, MD, PHD, Principal Investigator — Department of Oncology, Copenhagen University Hospital, Herlev, Herlev Ringvej 75, DK-2730 Herlev, Denmark
Locations (1):
- Department of Oncology, Copenhagen University Hospital, Herlev, Herlev, Denmark

REFERENCES:
- [Background] Svane IM, Pedersen AE, Johnsen HE, Nielsen D, Kamby C, Gaarsdal E, Nikolajsen K, Buus S, Claesson MH. Vaccination with p53-peptide-pulsed dendritic cells, of patients with advanced breast cancer: report from a phase I study. Cancer Immunol Immunother. 2004 Jul;53(7):633-41. doi: 10.1007/s00262-003-0493-5. Epub 2004 Feb 25. PMID 14985857